CLINICAL TRIAL: NCT07233980
Title: Therapist-Guided Internet-Delivered Cognitive Behaviour Therapy (CBT) for Chronic Conditions (Chronic Conditions Course; CCC): Single-Group Predictors of Change in Routine Care
Brief Title: Therapist-Guided Internet-Delivered CBT for Chronic Conditions: Predictors of Change
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Macquarie University, Australia (Other); Government of Saskatchewan, Ministry of Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-045b
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Physical Health Conditions
Keywords: Internet-delivered cognitive behavior therapy; Anxiety; Depression; Chronic physical health conditions; Therapist assistance; Predictors
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic Health Conditions Course_Therapist Guided ICBT (Experimental): All clients eligible for ICBT who report having a chronic health condition will receive the Wellbeing for Chronic Health Conditions Course. The course consists of 5 ICBT lessons released gradually over 8 weeks. Clients will also receive weekly support via secure messaging from a trained therapist for the duration of the course.
  Interventions: Behavioral: Internet-delivered CBT - Chronic Conditions Course (CCC)

INTERVENTIONS:
Behavioral: Internet-delivered CBT - Chronic Conditions Course (CCC) — The Wellbeing Course for Chronic Health Conditions is a transdiagnostic, internet-delivered cognitive behavioral intervention developed at Macquarie University. It is designed to help people living with chronic health conditions develop skills and strategies to maintain quality of life and emotional wellbeing. The course comprises 5 core online lessons released gradually over 8 weeks, targeting symptom identification, challenging unhelpful thoughts, pleasant activity scheduling, activity pacing and graded exposure, and relapse prevention. Each lesson is accompanied by downloadable exercise worksheets, case stories, and additional resources addressing challenges that clients may face alongside their chronic health conditions, such as assertive communication. Lesson materials are presented in a didactic, text-based format with visual supports. Therapists spend approximately 15 minutes each week responding to clients' messages and providing support.

SUMMARY:
Chronic health conditions are common, disabling, and often co-occur with depression and anxiety. Internet-delivered cognitive behaviour therapy (ICBT) reduces barriers to treatment and has been adapted for chronic conditions. A transdiagnostic approach is promising because it is both effective and convenient in that clients with diverse conditions receive the same program. Both therapist-guided and self-guided formats have been found effective; however, in routine care therapist support is most common to ensure that clients have support to personalize care.

This study evaluates the therapist-guided Chronic Conditions Course (CCC) and examines predictors of change. Past research shows that the most robust predictors of ICBT outcomes are baseline severity, adherence, credibility, and working alliance. However, few studies of ICBT for chronic conditions have examined predictors together. Moreover, the researchers are aware of no studies that have examined these core predictors in routine delivery of ICBT for those with chronic health conditions alongside other predictors-such as changes in thoughts and adaptive actions. A limitation of past work is that predictor analyses were typically secondary to trials designed for other purposes. This study directly addresses that gap by prospectively modeling predictors of change in routine care.

DETAILED DESCRIPTION:
The CCC is well supported by prior research. Dear and colleagues have completed several large trials validating the effectiveness of the CCC in addressing chronic health conditions. In the first large Randomized Controlled Trial (RCT; N=676), the researchers compared adults with diverse chronic conditions (e.g., multiple sclerosis, arthritis, epilepsy, diabetes, lupus, kidney disease, endometriosis, chronic pain, Parkinson's disease, chronic fatigue syndrome, COPD) when randomly assigned to the course compared to treatment as usual (Dear et al., 2022). Results showed significant improvements in depression, anxiety and disability versus treatment-as-usual, maintained at 12 months post-treatment. Effects were comparable to face-to-face care, requiring only ~10-20% of clinician time per patient. In a second large pragmatic RCT (N=850), with 24-month follow-up, preliminary results suggest clinically significant reductions in depression/anxiety, and improvements in disability and quality of life are maintained over time.

In Saskatchewan, the CCC is now offered as routine care (no cost) via the Online Therapy Unit (OTU). An RCT (N=178) by the team comparing therapist-guided (offered by a team of registered therapists based on scheduling) versus self-directed CCC found similar satisfaction, completion, and outcomes across formats. Most recently in a subsequent routine care sample (N=121) clients were found to make significant improvement in adaptive actions during treatment, but the study did not allow for comparison of the role or adaptive behaviours in predicting outcomes relative to other variables. The current study is a single-arm interventional trial designed to investigate predictors of outcome (primary outcomes are depression and anxiety). Variables of interest include baseline symptom severity, adherence, credibility, working alliance, adaptive actions, and therapeutic realizations controlling for demographic variables.

ELIGIBILITY:
Inclusion Criteria:

* Saskatchewan resident (as funding is provided by Saskatchewan government);
* Aged 18 years or older;
* self-reported diagnosed with chronic physical health condition affecting mental health;
* Access to a computer and the Internet;
* Consent to treatment/research

Exclusion Criteria:

* Current severe psychiatric or medical condition that requires immediate treatment and or would interfere with participation (e.g. current mania or psychosis, actively suicidal or unable to keep themselves safe, medical condition requiring immediate surgery or other invasive treatment, cognitive difficulties);
* Taking part in another treatment in our clinic;
* Living outside of Saskatchewan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Depression | Baseline (Screening), weeks 1-8, and 20 from enrollment
  Patient Health Questionnaire-9 (PHQ-9). Tracking the change in depression symptoms. 9 items are measured on a 4-point Likert scale ranging from 0-3. Scores are summed with total scores ranging from 0 to 27. Higher scores are associated with higher depression severity.
Anxiety | Baseline (Screening), weeks 1-8 and 20 from enrollment
  Generalized Anxiety Disorder-7 (GAD-7). Tracking the change in anxiety symptoms. 7 items are measured on a 4-point Likert scale ranging from 0-3. Scores are summed into a total score ranging from 0 to 21, with higher scores indicating more severe self-reported levels of anxiety.

SECONDARY OUTCOMES:
Average Pain Severity | Baseline (Screening), week 8 and week 20 from enrollment
  Visual Analogue Scale-Pain (VAS-Pain). The VAS-pain is a 3-item scale assessing pain experienced in the past 7-days. Items are rated on a line scale ranging from 0-10, and scores are summed into a total score ranging from 0-30. Higher scores indicate greater pain severity.
Functional Impairment | Baseline (Screening), weeks 4, 8, and 20 from enrollment
  Work and Social Adjustment Scale (WSAS). The WSAS is a measure of functional impairment experienced in different interpersonal and intrapersonal domains due to mental and physical health challenges. It includes 5 items rated on a 9-point Likert scale ranging from 0-8. Scores are summed to produce a total score between 0-40. Higher scores indicate greater impairment in functioning.
Treatment Satisfaction | Week 8
  Treatment Satisfaction Questionnaire (TSQ). A 13-item questionnaire used to assess satisfaction with treatment and negative effects experienced by clients during treatment. The questionnaire uses a combination of Likert scale [5-point (0-4) and 6-point (0-5)], open-ended, and dichotomous yes/no response options to gauge participants' perceptions of the course. The questionnaire was developed by Macquarie University, and has been adapted for use by the OTU. A total score is not produced for this measure.

OTHER OUTCOMES:
Treatment Credibility/Expectancy | Baseline (Screening) and week 4
  Credibility and Expectancy Questionnaire (CEQ). Measures treatment credibility and expectancy using 6 items, with two subscales. First three items correspond to the credibility subscale and the following three items correspond to the expectancy subscale. Items are measured on 9-point Likert scale ranging from 1-9. Subscale scores range from 3 to 27. Higher scores in each subscale indicate greater treatment credibility or treatment expectancy respectively.
Engagement Metrics | Weeks 2 to 8
  Homework Reflection Questionnaire. A 5-item questionnaire assessing week-to-week experience in the course, with items inquiring about the lesson participants worked on; effort exerted towards skills; helpfulness of lessons; and client successes, challenges and experiences over the previous week. A combination of checklist, Likert scale [7-point (1-7)], and open-ended response options are used to gauge participants' participation. The questionnaire is used by clinicians to monitor treatment. No overall score is produced.
Working Alliance | Week 4
  Working Alliance Inventory for Guided Internet Interventions (WAI-I). The WAI-I is a 12-item measure assessing therapist-client alliance and client-program alliance. Items are measured on a 5-point Likert scale ranging from 1-5, and scores are summed to produce a total score ranging from 12 to 60. Higher scores on this scale indicate higher levels of client-program alliance and therapist-client alliance.
Adaptive Actions | Baseline (Screening), weeks 4, 8, and 20 post enrollment
  Things You Do Questionnaire-15 (TYDQ-15). A measure of behaviors associated with mental health. 15 items are measured on a 5-point Likert scale ranging from 0-4. Subscales include Healthy Routine, Healthy Thinking, Social Connection, Meaningful Activities, and Goals and Plans. Scores are summed into subscale scores ranging from 0 to 12, and a total score ranging from 0 to 60, with higher scores indicating increased engagement in behaviours associated with mental health.
Therapeutic Realization | Baseline(Screening), weeks 4, 8, and 20 from enrollment
  Demoralization and Insight Scale (DIS). The DIS is a 9-item revised version of the Therapeutic Realization Scale-revised, used to assess the extent to which clients feels less demoralized and gain insight during treatment. Items on this scale are measured on a 4-point Likert scale ranging from 0-3, and scores are summed to produce a total score ranging from 0-27. Higher scores indicate higher therapeutic realization.
Treatment Adherence | Calculated at Week 8
  The Online Therapy Unit system collects information on the number of lessons completed, and number of emails client exchange with their therapist. Clients' adherence to treatment is calculated by averaging the sum of all lessons completed, all emails sent and all emails received from therapists.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (2):
- Canada (2):
  - Online Therapy Unit, University of Regina, Regina, Saskatchewan
  - Online Therapy Unit, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zalaznik D, Strauss AY, Halaj A, Barzilay S, Fradkin I, Katz BA, Ganor T, Ebert DD, Andersson G, Huppert JD. Patient alliance with the program predicts treatment outcomes whereas alliance with the therapist predicts adherence in internet-based therapy for panic disorder. Psychother Res. 2021 Nov;31(8):1022-1035. doi: 10.1080/10503307.2021.1882712. Epub 2021 Feb 10. PMID 33567994
- [Background] Dear BF, Scott AJ, Fogliati R, Gandy M, Karin E, Dudeney J, Nielssen O, McDonald S, Heriseanu AI, Bisby MA, Sharpe L, Jones MP, Ali S, Titov N. The Chronic Conditions Course: A Randomised Controlled Trial of an Internet-Delivered Transdiagnostic Psychological Intervention for People with Chronic Health Conditions. Psychother Psychosom. 2022;91(4):265-276. doi: 10.1159/000522530. Epub 2022 Apr 1. PMID 35367986
- [Background] Mehta SH, Nugent M, Peynenburg V, Thiessen D, La Posta G, Titov N, Dear BF, Hadjistavropoulos HD. Internet-delivered cognitive behaviour therapy for chronic health conditions: self-guided versus team-guided. J Behav Med. 2022 Oct;45(5):674-689. doi: 10.1007/s10865-022-00346-x. Epub 2022 Aug 3. PMID 35921055
- See also: Trial registration of the second large pragmatic RCT — https://www.anzctr.org.au/Trial/Registration/TrialReview.aspx?ACTRN=12620000969965